CLINICAL TRIAL: NCT06371248
Title: Steady Feet Falls Prevention Programme for Community-dwelling Older Adults at Risk for Falls in Singapore: A Feasibility Study
Brief Title: Steady Feet: Preventing Falls in the Community
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Changi General Hospital (Other)
Responsible Party: Principal Investigator, Low Shou Lin, Principal Investigator, Changi General Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2850
Record Dates: First submitted 2024-04-08; First posted 2024-04-17 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Fall; Feasibility; Older Adults; Exercise
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Three-month, twice weekly, exercise intervention and usual care for fall prevention.
  Interventions: Behavioral: Steady Feet; Other: Usual care for fall prevention
- Control (Active Comparator): Usual care for fall prevention.
  Interventions: Other: Usual care for fall prevention

INTERVENTIONS:
Behavioral: Steady Feet — Steady Feet is a three-month progressive exercise-based single-component intervention spanning twenty-four sessions, with a focus on enhancing balance, mobility, and strength among community-dwelling older adults at risk of falls.
  Arms: Intervention
Other: Usual care for fall prevention — CGH's usual care for fall prevention, which include fall prevention materials and advice.

SUMMARY:
The purpose of this study is to examine the feasibility of Steady Feet, a three-month community-based falls prevention exercise program.

DETAILED DESCRIPTION:
Participants aged 60 or older, at high risk of falls, with Short Physical Performance Battery (SPPB) scores between 7 and 11, and without significant cognitive or vision impairment, were recruited for a non-randomized, two-arm study. They were evaluated at baseline and the third month. The intervention group (IG) underwent Steady Feet and CGH's standard care for fall prevention, while the control group (CG) received CGH's standard care for fall prevention. Feasibility was assessed across Bowen's domains, including acceptability, demand, implementation, practicality, adaptation, and limited efficacy. Measurements included SPPB, Timed Up and Go, the 6-minute walk test, the Four-Square Step Test, the CONFbal scale, and a satisfaction survey administered to IG participants. Between-groups statistical analyses will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Aged 60 years and above
* At high risk of falls according to the FROP-COM
* Short Physical Performance Battery (SPPB) score of 7 to 11
* Able to ambulate without wheelchairs or walkers
* Able to understand basic instructions.

Exclusion Criteria:

* Possess significant cognitive impairment (Abbreviated Mental Test < 5)
* Had visual impairment, as determined by not passing at least 2 out of 3 Vision Function Test(s) (Logarithm of the Minimum Angle of Resolution (LogMar) vision, Stereoscopic vision, and Melbourne Edge Test (MET)

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2018-11-19 (Actual); Primary Completion 2019-12-20 (Actual); Study Completion 2019-12-20 (Actual)

PRIMARY OUTCOMES:
Short Physical Performance Battery (SPPB) | an average of 12 weeks
  SPPB comprises three components, (i) static balance, (ii) gait speed, and (iii) chair stands. A higher score on the SPPB is indicative of better physical functional status (maximum score of 12 points).

SECONDARY OUTCOMES:
CONFbal | an average of 12 weeks
  The CONFbal scale is a ten-item measure used to assess self-reported confidence in maintaining balance under different conditions. The overall CONFbal score ranges from 10 to 30. Lower scores reflect higher levels of subjective balance confidence.
Six-minute walk test (6MWT) | an average of 12 weeks
  The 6MWT is a validated tool for assessing functional status and endurance in older adults. Participants are instructed to walk continuously for six minutes along a ten-meter course, which is marked with a turnaround point to enable participants to walk to-and-fro. The total distance walked during the test is recorded.
Timed up and go (TUG) | an average of 12 weeks
  The TUG is used to evaluate gait, balance, and dynamic mobility in individuals. Participants are instructed to rise from a seated position, walk three meters to the endpoint marked with an object, and return to the seat. The time taken to complete the assessment is recorded.
Four square step test (FSST) | an average of 12 weeks
  The FSST is a validated measure of coordination and dynamic stability in older adults. Participants are asked to quickly step forward, backward, and sideways over a low obstacle, following a predetermined sequence delineated by four squares marked on the ground. The time taken to complete the task was recorded.
Feedback and satisfaction survey | an average of 12 weeks
  The self-developed feedback and satisfaction survey assessed participant satisfaction with the SF sessions, the instructors, the venue, the pace, the exercises, and the perceived effects of SF on their health

OTHER OUTCOMES:
Attendance and completion rates | an average of 12 weeks
  Participants' attendance and completion records for the Steady Feet intervention.
Safety of Steady Feet | an average of 12 weeks
  Reports on adverse events (if any) during the study.

CONTACTS AND LOCATIONS:
Overall Officials: Shou Lin Low, MRCP (UK), Principal Investigator — Changi General Hospital
Locations (1):
- Changi General Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No
The data that support the findings of this study are available on request from the corresponding author. The data are not publicly available due to ethical restrictions.